CLINICAL TRIAL: NCT06141512
Title: Improvements in Aerobic Fitness With Exercise Training: the Role of Myokines
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stirling (Other)
Responsible Party: Principal Investigator, Niels Vollaard, Principal Investigator, University of Stirling
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UStirling
Record Dates: First submitted 2023-11-13; First posted 2023-11-21 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: General Health
Keywords: VO2max; Myokine; Cardiorespiratory Fitness
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: All participants will undergo the same exercise training intervention. Based on the outcome measure of VO2max, participants will be divided into groups with a low response for VO2max, a medium response, and a high response for VO2max. It will be investigated whether the change in plasma myokine levels differs between the 3 groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reduced-exertion high-intensity interval training (REHIT) (Experimental): All participants complete 6 weeks (3 sessions/week) of an exercise intervention labelled 'REHIT'.
  Exercise sessions involve 10 minutes of unloaded cycling interspersed with 2 x 20 sec 'all-out' sprints against a resistance of 7.5% of participant's body weight. Sprints begin at 1:40 min and 5:40 min.
  Interventions: Behavioral: Reduced-exertion high-intensity interval training (REHIT)

INTERVENTIONS:
Behavioral: Reduced-exertion high-intensity interval training (REHIT) — Description same as Arm description.
  Other Names: Sprint interval training (SIT)

SUMMARY:
For both healthy adults and patients with cardiovascular disease (CVD), aerobic fitness (V̇O2max) is a stronger predictor of the risk of future chronic disease and premature death than other established risk factors such as hypertension, smoking, or Type 2 diabetes. It is important to improve the understanding of the regulation of V̇O2max to enable optimisation of interventions aimed at increasing V̇O2max in the current predominantly sedentary population. Currently, only exercise training is a viable method for increasing V̇O2max. However, ~10-20% of people who follow fully supervised, standardised training interventions do not demonstrate a measurable increase in V̇O2max. Low response to training is a clinically relevant concern, but the large variability in response to exercise training also provides an opportunity to dissect out the molecular mechanisms responsible for adaptations to V̇O2max by contrasting low vs. high responders to training. It has been previously demonstrated that low responders for VO2max fail to up regulate a number of genes that encode putative 'myokines', while the high responders demonstrated a significant increase in the expression of these genes, suggesting these myokines may play an important mechanistic role in modulating VO2max. The aim of the present study is to examine whether low responders for VO2max have an attenuated increase in the plasma levels of the previously identified myokines.

DETAILED DESCRIPTION:
For both healthy adults and patients with cardiovascular disease (CVD), aerobic fitness (V̇O2max) is a stronger predictor of the risk of future chronic disease and premature death than other established risk factors such as hypertension, smoking, or Type 2 diabetes. Considering the large medical and economic burden of physical inactivity-related chronic disease it is important to improve the understanding of the regulation of V̇O2max to enable optimisation of interventions aimed at increasing V̇O2max in the current predominantly sedentary population. Furthermore, there is a need to identify novel drug targets to aid pharmacological intervention in those individuals who are unwilling or unable to improve V̇O2max through exercise.

Currently, only exercise training is a viable method for increasing V̇O2max. However, although exercise training on average improves V̇O2max, ~10-20% of people who follow fully supervised, standardised training interventions do not demonstrate a measurable increase in V̇O2max. Low response to training is a clinically relevant concern, but the large variability in response to exercise training also provides an opportunity to dissect out the molecular mechanisms responsible for adaptations to V̇O2max by contrasting low vs. high responders to training.

Using this approach it has previously been shown that in skeletal muscle samples obtained pre- and post- training, 86 genes are differentially regulated in high compared to low responders for V̇O2max. Strikingly, out of these 86 genes, 13 genes encode proteins that have been reported to be released by muscle during or after exercise (i.e., 'messenger proteins' termed myokines). This strongly suggests low responders to exercise training fail to sufficiently upregulate the production and release of these myokines, and that this is (at least partly) the reason why these people do not manage to improve their V̇O2max as much as high responders. However, in order to confirm a mechanistic role of these myokines in increasing V̇O2max, it needs to be demonstrated that beside the change in gene expression, the change in the plasma levels of these myokines is also impaired in low responders for V̇O2max.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age ≥ 18 y or <40 y
* BMI < 35 kg/m2
* otherwise healthy, untrained individuals

Exclusion Criteria:

* Age <18 y or >40 y
* BMI > 35 kg/m2
* classification of 'highly physically active' according to the International Physical Activity Questionnaire (IPAQ)
* answering 'yes' to one or more questions on a standard Physical Activity Readiness Questionnaire (PAR-Q)
* resting heart rate ≥100bpm, clinically significant hypertension (140/90 mmHg)
* a personal history of metabolic or cardiovascular disease
* Female participants because of unknown effects of the menstrual cycle on the levels of the measured myokines.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Training induced changes in VO2max | Pre-intervention and 3 days post-intervention
  Maximal aerobic capacity (VO2max) will be measured pre- and post-training to determine the change in VO2max.
Training induced changes in plasma myokines | Pre-intervention and 3 days post-intervention
  Plasma myokine levels of 8 myokines will be measured pre- and post-training to determine the change in plasma myokine levels.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Vollaard, PhD, Principal Investigator — University of Stirling
Locations (1):
- University of Stirling, Stirling, United Kingdom

IPD SHARING:
Plan to Share IPD: No